CLINICAL TRIAL: NCT03944694
Title: White Cell Ratios as Markers of Delirium and Outcome in Acute Ischemic Stroke. DELirium in Acute Ischemic Stroke [DELIAS]
Brief Title: White Cell Ratios as Markers of Delirium and Outcome in Acute Ischemic Stroke.
Acronym: DELIAS
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Katarzyna Kotfis, Principal Investigator, Pomeranian Medical University Szczecin
Other Study IDs: 0012/84/03/19
Record Dates: First submitted 2019-05-08; First posted 2019-05-09 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Delirium; Ischemic Stroke
Keywords: delirium; stroke; neutrophil-to-lymphocyte ratio; NLR; mortality
MeSH Terms: conditions — Delirium; Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirious: Patients were delirious if CAM-ICU was positive within 24 hours from admission due to acute ischemic stroke.
  Interventions: Diagnostic Test: Delirium assessment.
- Non-delirious: Patients were delirious if CAM-ICU was negative within 24 hours from admission due to acute ischemic stroke.
  Interventions: Diagnostic Test: Delirium assessment.

INTERVENTIONS:
Diagnostic Test: Delirium assessment. — Full blood count analysis.

SUMMARY:
The aim of this study was to investigate the role of Neutrophil-to-Lymphocyte Ratio (NLR) and other derived white cell markers as early markers of delirium and outcome after acute ischemic stroke (AIS).

DETAILED DESCRIPTION:
Delirium is an acute brain disorder, potentially reversible, commonly occurring in patients with acute ischemic stroke. The pathomechanism of delirium is related to neuroinflammatory process and oxidative stress. Search for readily available diagnostic marker that will aid clinicians in early identification of delirium is an on-going process. The aim of this study was to investigate the role of Neutrophil-to-Lymphocyte Ratio (NLR) and other derived white cell markers as early markers of delirium and outcome after acute ischemic stroke (AIS).

ELIGIBILITY:
Inclusion Criteria:

* age >18 years)
* acute ischemic stroke

Exclusion Criteria:

* hematology disorders
* incomplete laboratory testing
* no data regarding follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients (age >18 years) with acute ischemic stroke, admitted to a neurology department of a busy district general hospital in Poland between 30.06.2015 and 31.03.2018. Patients with AIS were admitted to the neurology department within 48 hours of symptom development.
Sampling Method: Non-Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2015-06-30 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Early-onset-delirium. | 24 hours
  Delirium within 24 hours from admission.

SECONDARY OUTCOMES:
Mortality at 30 days. | 30 days
  Mortality determined at follow-up on day 30 after acute ischemic stroke.
Mortality at 1 year. | 1 year
  Mortality determined at follow-up at 1 year after acute ischemic stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Rotter, MD, PhD, Study Chair — Pomeranian Medical University Szczecin

IPD SHARING:
Plan to Share IPD: No